CLINICAL TRIAL: NCT00269490
Title: Yoga as an Adjunctive Therapy for Post-Traumatic Stress Disorder: A Feasibility Study
Brief Title: Yoga as a Therapy for Traumatic Experiences
Status: Completed | Type: Observational
Sponsor: Samueli Institute for Information Biology (Other)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Other Study IDs: WU# 05-89014; DoD Assurance No. P60001; FWA #00001628; USU IRB Reference G188JO
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post-Traumatic Stress Disorder; Yoga Nidra
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Yoga Nidra

SUMMARY:
The purpose of the proposed research is to conduct a feasibility study of yoga as an adjunctive therapy for the treatment of posttraumatic stress disorder (PTSD) in 15 military personnel at the Walter Reed Army Medical Center (WRAMC) in Washington, DC. Participants will complete 10 weeks of yoga training, in addition to the continuing their usual and customary care for PTSD at WRAMC. The style of yoga chosen for this study, Yoga Nidra, uses deep relaxation, deep breathing and meditation to systematically reduce physical, emotional, mental, and even subconscious tension. After a diagnostic mental health assessment at baseline, participants will attend a total of 18 classes taught over a 10-week period and will practice daily at home using a compact disk provided by the instructor. Baseline measures will include the Patient Health Questionnaire, PD-HAT Trauma Questions, PTSD Symptom Scale - Interview, Fear of Loss of Vigilance Scale, and expectation of efficacy. The primary outcome measure will be the PTSD Checklist. Changes in health status, locus of control, and pain will be assessed over the course of the study. An additional goal of this study is to gather preliminary data on the anticipated effect size and feasibility of conducting a larger clinical study of the adjunctive use of yoga for the treatment of PTSD symptoms in enlisted military personnel.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty military personnel
* Aged 18 and over
* A minimum score of 40 on the Posttraumatic Stress Disorder Checklist (PCL-M), a brief, self-report instrument used to assess PTSD severity.

Exclusion Criteria:

* Active suicidal or homicidal ideation
* Severe cognitive impairment or history of cognitive disorder
* Serious surgical procedures within the last two months or planned
* Treatment for refractory pain
* New or dose adjusted psychotropic medication (i.e. SSRIs and anxiolytics) in last month
* Unwilling or unable to practice Yoga Nidra at home
* Amputation of any body part

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-12; Primary Completion 2006-10 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: COL Charles C Engel, MD, MPA, Principal Investigator — Walter Reed Army Medical Center; Christine Goertz Choate, DC, PhD, Principal Investigator — Samueli Institute for Information Biology
Locations (1):
- Deployment Health Clinical Center, Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States